CLINICAL TRIAL: NCT03491956
Title: Double Filtration Plasmapheresis (DFPP) Improves Lipid Profile and Platelet Function in Hyperlipidemia Patients
Brief Title: Double Filtration Plasmapheresis (DFPP) and Lipid Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pudong Hospital (Other)
Responsible Party: Principal Investigator, Jin HM, MD, Professor, Shanghai Pudong Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiPudongH2
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: DFPP and Platelet Function

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DFPP group (Other): self contrast (before and after DFPP)
  Interventions: Device: DFPP

INTERVENTIONS:
Device: DFPP — Lipid levels,platelet function，and platelet RNA sequencing in hyperlipidemia patients before and after DFPP

SUMMARY:
Little clinic trials showed that Double Filtration Plasmapheresis (DFPP) could improve lipid metabolism, however, whether DFPP can improve platelet function and recover Endothelial function is unknown. In this study, we try to confirm the hypothesis that DFPP can improve endothelial function in hyperlipidemia patients.

ELIGIBILITY:
Inclusion Criteria:

1. hyperlipidemia

Exclusion Criteria:

1. Severe liver and kidney dysfunction
2. Severe cardiopulmonary insufficiency
3. tumor
4. pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
lipid levels | 1 year
  reduce in lipid levels

SECONDARY OUTCOMES:
Platelet RNA sequencing | 1 year
  whether the RNA sequencing of platelet changed ?

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, doctor, Principal Investigator — Shanghai Pudong Hospital
Locations (1):
- Shanghai Pudong Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang XM, Gu YH, Deng H, Xu ZQ, Zhong ZY, Lyu XJ, Jin HM, Yang XH. Plasma Purification Treatment Relieves the Damage of Hyperlipidemia to PBMCs. Front Cardiovasc Med. 2021 Jul 7;8:691336. doi: 10.3389/fcvm.2021.691336. eCollection 2021. PMID 34307504